CLINICAL TRIAL: NCT02488967
Title: A Randomized Phase III Trial of Adjuvant Therapy Comparing Doxorubicin Plus Cyclophosphamide Followed by Weekly Paclitaxel With or Without Carboplatin for Node-Positive or High-Risk Node-Negative Triple-Negative Invasive Breast Cancer
Brief Title: Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel With or Without Carboplatin in Treating Patients With Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BR003; NCI-2015-00128 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BR1428; NRG-BR003 (Other: NRG Oncology); NRG-BR003 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Breast Adenocarcinoma; Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor Negative; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIC Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (AC-->WP) (Active Comparator): Patients receive doxorubicin hydrochloride IV over 15 minutes and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive paclitaxel IV over 60 minutes on day 1. Treatment repeats weekly for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm II (AC-->WP + carboplatin) (Experimental): Patients receive doxorubicin hydrochloride and cyclophosphamide as in Arm I. Patients then receive paclitaxel IV over 60 minutes on days 1, 8, and 15 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II (AC-->WP + carboplatin)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This randomized phase III trial studies how well doxorubicin hydrochloride and cyclophosphamide followed by paclitaxel with or without carboplatin work in treating patients with triple-negative breast cancer. Drugs used in chemotherapy, such as doxorubicin hydrochloride, cyclophosphamide, paclitaxel, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether doxorubicin hydrochloride and cyclophosphamide is more effective when followed by paclitaxel alone or paclitaxel and carboplatin in treating triple-negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of carboplatin to an adjuvant chemotherapy regimen of doxorubicin (doxorubicin hydrochloride)/cyclophosphamide followed by paclitaxel will improve the invasive disease-free survival (IDFS) compared to doxorubicin/cyclophosphamide followed by paclitaxel when administered to patients with operable node-positive or high-risk node-negative triple-negative breast cancer.

SECONDARY OBJECTIVES:

I. To determine whether the addition of carboplatin to an adjuvant chemotherapy regimen of doxorubicin/cyclophosphamide followed by paclitaxel will improve the overall survival (OS) compared to doxorubicin/cyclophosphamide followed by paclitaxel when administered to patients with operable node-positive or high-risk node-negative triple-negative breast cancer.

II. To determine whether the addition of carboplatin to an adjuvant chemotherapy regimen of doxorubicin/cyclophosphamide followed by paclitaxel will improve the breast cancer-free survival (BCFS) compared to doxorubicin/cyclophosphamide followed by paclitaxel when administered to patients with operable node-positive or high-risk node-negative triple-negative breast cancer.

III. To determine whether the addition of carboplatin to an adjuvant chemotherapy regimen of doxorubicin/cyclophosphamide followed by paclitaxel will improve the recurrence-free interval (RFI) compared to doxorubicin/cyclophosphamide followed by paclitaxel when administered to patients with operable node-positive or high-risk node-negative triple-negative breast cancer.

IV. To determine whether the addition of carboplatin to an adjuvant chemotherapy regimen of doxorubicin/cyclophosphamide followed by paclitaxel will improve the distant recurrence-free interval (DRFI) compared to doxorubicin/cyclophosphamide followed by paclitaxel when administered to patients with operable node-positive or high-risk node-negative triple-negative breast cancer.

V. To determine the toxicity of doxorubicin/cyclophosphamide followed by paclitaxel administered concurrently with carboplatin compared to the toxicity of doxorubicin/cyclophosphamide followed by paclitaxel alone.

VI. To determine if germline breast cancer (BRCA) status is associated with benefit in IDFS or OS from the addition of carboplatin to an adjuvant chemotherapy regimen of doxorubicin/cyclophosphamide followed by paclitaxel in patients with operable node-positive or high-risk node-negative triple-negative breast cancer.

VII. To determine if the addition of carboplatin will improve the RFI among the homologous recombination (HR) deficient patients as determined by the homologous recombination deficiency (HRD) score.

VIII. To determine whether the efficacy of carboplatin on RFI in HR-deficient patients differs from that in patients who are not HR-deficient.

IX. To collect tissue and blood samples at several occasions for future biomarkers development in predicting risk of breast cancer recurrence in patients with operable node-positive or high-risk node-negative triple-negative breast cancer treated with doxorubicin/cyclophosphamide followed by paclitaxel with or without carboplatin and predicting benefit from the addition of carboplatin among these patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (DOXORUBICIN HYDROCHLORIDE [A] CYCLOPHOSPHAMIDE [C]-->WEEKLY PACLITAXEL [WP]): Patients receive doxorubicin hydrochloride intravenously (IV) over 15 minutes and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive paclitaxel IV over 60 minutes on day 1. Treatment repeats weekly for 12 courses in the absence of disease progression or unacceptable toxicity.

ARM II (AC-->WP + CARBOPLATIN): Patients receive doxorubicin hydrochloride and cyclophosphamide as in Arm I. Patients then receive paclitaxel IV over 60 minutes on days 1, 8, and 15 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 5 years and then every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed and dated an institutional review board (IRB)-approved consent form that conforms to federal and institutional guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* The tumor must be unilateral invasive adenocarcinoma of the breast on histologic examination
* All of the following staging criteria (according to the 7th edition of the American Joint Committee on Cancer [AJCC] Cancer Staging Manual) must be met:

  * By pathologic evaluation, primary tumor must be pT1-3
  * By pathologic evaluation, ipsilateral nodes must be pN0, pN1 (pN1mi, pN1a, pN1b, pN1c), pN2a, pN2b, pN3a, or pN3b
  * If pN0, pathological tumor must be greater than or equal to 3.0 cm
* The tumor must have been determined to be human epidermal growth factor receptor 2 (HER2)-negative as follows:

  * Immunohistochemistry (IHC) 0-1+; or
  * IHC 2+ and in situ hybridization (ISH) non-amplified with a ratio of HER2 to centromere enumerator probe 17 (CEP17) less than 2.0, and if reported, average HER2 gene copy number less than 4 signals/cells; or
  * ISH non-amplified with a ratio of HER2 to CEP17 less than 2.0, and if reported, average HER2 gene copy number less than 4 signals/cells
* The tumor must have estrogen receptor (ER)-and progesterone receptor (PgR)-status assessed using current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines; patients are eligible if the tumor staining meets one of the following criteria:
* ER-negative and PgR-negative by ASCO/CAP guidelines, OR
* ER or PgR stains are positive in 1-9% of cells and neither is positive in greater than or equal to 10% of cells.
* The patient must have undergone either a mastectomy (total, skin-sparing, or nipple-sparing) or lumpectomy
* For patients who undergo lumpectomy, the margins of the resected specimen must be histologically free of invasive tumor and ductal carcinoma in situ (DCIS) as determined by the local pathologist; if pathologic examination demonstrates tumor at the line of resection, additional excisions may be performed to obtain clear margins; if tumor is still present at the resected margin after re-excision(s), the patient must undergo mastectomy to be eligible; (patients with margins positive for lobular carcinoma in situ [LCIS] are eligible without additional resection)
* For patients who undergo mastectomy, the margins must be free of residual gross tumor; (patients with microscopic positive margins are eligible as long as post-mastectomy radiation therapy [RT] of the chest wall will be administered)
* The patient must have completed one of the procedures for evaluation of pathologic nodal status listed below.

  * Sentinel lymphadenectomy alone:

    * If pathologic nodal staging based on sentinel lymphadenectomy is pN0 or pN1b;
    * If pathologic nodal staging based on sentinel lymphadenectomy is pN1mi or pN1a and the patient has undergone breast conserving surgery (with planned breast radiotherapy), the primary tumor must be T1 or T2 by pathologic evaluation and the nodal involvement must be limited to 1 or 2 positive nodes
  * Sentinel lymphadenectomy followed by removal of additional non-sentinel lymph nodes if the sentinel node (SN) is positive; or
  * Axillary lymphadenectomy with or without SN isolation procedure
* The interval between the last surgery for breast cancer (including re-excision of margins) and randomization must be no more than 60 days
* Absolute neutrophil count (ANC) must be greater than or equal to1200/mm^3
* Platelet count must be greater than or equal 100,000/mm^3
* Hemoglobin must be greater than or equal to 10 g/dL
* Adequate hepatic function must be met based on the results of the most recent postoperative tests performed with 6 weeks prior to randomization.
* Total bilirubin must be less than or equal to upper limit of normal (ULN) for the laboratory (lab) unless the patient has a bilirubin elevation greater than ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin
* Alkaline phosphatase must be less than or equal to 2.5 x ULN for the lab
* Aspartate aminotransferase (AST) must be less than or equal to 1.5 x ULN for the lab

  * Note: If alanine aminotransferase (ALT) is performed instead of AST (per institution's standard practice), the ALT value must be less than or equal to 1.5 x ULN; if both were performed, the AST must be less than or equal to 1.5 x ULN.
* Patients with AST or alkaline phosphatase greater than ULN are eligible for inclusion in the study if liver imaging (computed tomography [CT], magnetic resonance imaging [MRI], positron emission tomography [PET]-CT, or PET scan) performed within 90 days prior to randomization does not demonstrate metastatic disease and the requirements above are met
* Patients with alkaline phosphatase that is greater than ULN but less than or equal to 2.5 x ULN or unexplained bone pain are eligible for inclusion in the study if a bone scan, PET-CT scan, or PET scan performed within 90 days prior to randomization does not demonstrate metastatic disease
* Adequate renal function determined within 6 weeks prior to randomization defined as the most recent serum creatinine less than or equal to ULN or measured or calculated creatinine clearance greater than 60 mL/min
* Left ventricular ejection fraction (LVEF) assessment must be performed within 90 days prior to randomization; (LVEF assessment performed by 2-dimensional [D] echocardiogram is preferred; however, multi gated acquisition [MUGA] scan may be substituted based on institutional preferences;) the LVEF must be greater than or equal to 50% regardless of the cardiac imaging facility's lower limit of normal.

Exclusion Criteria:

* T4 tumors including inflammatory breast cancer
* Definitive clinical or radiologic evidence of metastatic disease; required imaging studies must have been performed within 90 days prior to randomization
* Synchronous or previous contralateral invasive breast cancer; (patients with synchronous and/or previous contralateral DCIS or LCIS are eligible)
* Any previous history of ipsilateral invasive breast cancer or ipsilateral DCIS; (patients with synchronous or previous ipsilateral LCIS are eligible)
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior to randomization
* Previous therapy with anthracyclines or taxanes for any malignancy
* Chemotherapy administered for the currently diagnosed breast cancer prior to randomization
* Any continued use of sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy; patients are eligible if these medications are discontinued prior to randomization
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens; this includes but is not confined to:

  * Active cardiac disease

    * Angina pectoris that requires the current use of anti-anginal medication;
    * Ventricular arrhythmias except for benign premature ventricular contractions;
    * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication;
    * Conduction abnormality requiring a pacemaker;
    * Valvular disease with documented compromise in cardiac function; or
    * Symptomatic pericarditis
  * History of cardiac disease

    * Myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricle (LV) function;
    * History of documented congestive heart failure (CHF); or
    * Documented cardiomyopathy
* Uncontrolled hypertension defined as sustained systolic blood pressure (BP) greater than 150 mmHg or diastolic BP greater than 90 mmHg; (patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria)
* Active hepatitis B or hepatitis C with abnormal liver function tests
* Patients known to be human immunodeficiency virus (HIV) positive with a baseline cluster of differentiation (CD)4 count of less than 250 cells/mm^3 or have a history of acquired immune deficiency syndrome (AIDS) indicator conditions
* Intrinsic lung disease resulting in dyspnea
* History of hospitalization in past 12 months for diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemic nonketotic syndrome (HHNS)
* Active infection or chronic infection requiring chronic suppressive antibiotics
* Nervous system disorder (paresthesia, peripheral motor neuropathy, or peripheral sensory neuropathy) greater than or equal to grade 2, per the Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0
* Conditions that would prohibit administration of corticosteroids
* Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids)
* Known hypersensitivity to any of the study drugs or excipients, e.g., polysorbate 80 and Cremophor® EL
* Other non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements
* Pregnancy or lactation at the time of study entry; (note: pregnancy testing according to institutional standards for women of childbearing potential must be performed within 2 weeks prior to randomization)
* Use of any investigational product within 4 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Estimated)
Dates: Start 2015-07-26; Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
IDFS | Up to 10 years
  IDFS events are local invasive recurrence after mastectomy, local invasive recurrence in the ipsilateral breast after lumpectomy, regional recurrence, distant recurrence, contralateral invasive breast cancer, second non-breast primary cancer (excluding squamous or basal cell carcinoma of the skin), or death from any cause before recurrence or second primary cancer. IDFS will be compared between the two treatment arms by the stratified log-rank test. The Kaplan-Meier estimates will be calculated separately for patients under the different treatment regimens.

SECONDARY OUTCOMES:
BCFS | From randomization until local recurrence (invasive or DCIS), regional recurrence, or distant recurrence, contralateral breast cancer (invasive or DCIS), or death from any causes, assessed up to 10 years
  The stratified log-rank tests will be 2-sided with significance level 0.05. Treatment efficacy in these secondary endpoints will be assessed by Cox models adjusting for clinical factors such as age, number of positive nodes, BRCA mutation status, tumor size, and tumor grade.
DRFI | From randomization until distant metastasis or death from breast cancer, regardless of occurrence of any intervening local or regional recurrences, contralateral breast cancers, or non-breast second primary cancers, assessed up to 10 years
  The stratified log-rank tests will be 2-sided with significance level 0.05. Treatment efficacy in these secondary endpoints will be assessed by Cox models adjusting for clinical factors such as age, number of positive nodes, BRCA mutation status, tumor size, and tumor grade.
Frequencies of adverse events categorized using the National Cancer Institute CTCAE v4.0 | Up to 10 years
  Frequencies of all adverse events during the treatment period will be tabulated by treatment, toxicity type, and grade. The Pearson Chi-squared test with continuity adjustment will be used to compare toxicity grades in each type between the two treatment regimens. The test will be 2-sided with significance level 0.05.
OS | From randomization until death from any cause, assessed up to 10 years
  The stratified log-rank tests will be 2-sided with significance level 0.05. Treatment efficacy in these secondary endpoints will be assessed by Cox models adjusting for clinical factors such as age, number of positive nodes, BRCA mutation status, tumor size, and tumor grade.
RFI | From randomization until invasive local, regional, or distant recurrence, or death from breast cancer (censored for death from other causes), assessed up to 10 years
  The stratified log-rank tests will be 2-sided with significance level 0.05. Treatment efficacy in these secondary endpoints will be assessed by Cox models adjusting for clinical factors such as age, number of positive nodes, BRCA mutation status, tumor size, and tumor grade.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Valero, Principal Investigator — NRG Oncology
Locations (1296):
- United States (1286):
  - Southern Cancer Center PC-Mobile, Mobile, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Southern Cancer Center PC-Springhill, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Breast Cancer Specialists-Gilbert, Gilbert, Arizona
  - Virginia G Piper Cancer Care-Glendale, Glendale, Arizona
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Oncology Associates-Biltmore Cancer Center, Phoenix, Arizona
  - Arizona Breast Cancer Specialists-Phoenix, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Breast Cancer Specialists, Scottsdale, Arizona
  - Arizona Breast Cancer Specialists-Scottsdale, Scottsdale, Arizona
  - Oncogyne PC-Arizona Oncology, Scottsdale, Arizona
  - Virginia G Piper Cancer Care-Del Camino, Scottsdale, Arizona
  - Sedona Medical Center, Sedona, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Enloe Medical Center, Chico, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Dominican Santa Cruz Hospital, Santa Cruz, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Joseph's Medical Center, Stockton, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale-New Haven Shoreline Medical Center, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Lawrence and Memorial Cancer Center, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - AMITA Health Cancer Institute and Outpatient Center, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Genesis Cancer Center - Silvis, Silvis, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - The Community Hospital, Munster, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Saint Elizabeth Fort Thomas, Fort Thomas, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Norton Audubon Hospital and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - CHRISTUS Saint Patrick Hospital, Lake Charles, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - Mercy Hospital, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Kensington Medical Center, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Richard A Henson Cancer Institute at Ocean Pines, Ocean Pines, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Maryland Oncology Hematology PA-Aquilino Cancer Center, Rockville, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Bloomfield, Bloomfield, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital ? Dearborn, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - UP Health System Hematology Oncology Marquette, Marquette, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Highland Hospital, Rochester, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Randolph Hospital, Asheboro, North Carolina
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Rex Hematology Oncology Associates-Cary, Cary, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute-Tryon, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Levine Cancer Institute - Rutherford, Forest City, North Carolina
  - Rex Hematology Oncology Associates-Garner, Garner, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kenansville, Kenansville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Rex Hematology Oncology Associates-Blue Ridge, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Vidant Oncology-Richlands, Richlands, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Marion L Shepard Cancer Center at Vidant Beaufort Hospital, Washington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Compass Oncology East, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Compass Oncology West, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Compass Oncology Tualatin, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Suburban Community Hospital and Cancer Center, Norristown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - Texas Cancer Center, Abilene, Texas
  - Texas Oncology PA - Amarillo, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Texas Cancer Center - Medical City Dallas, Dallas, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Texas Tech University Health Sciences Center-El Paso, El Paso, Texas
  - Texas Oncology-El Paso, El Paso, Texas
  - Texas Oncology-Flower Mound, Flower Mound, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Oncology - Garland, Garland, Texas
  - Texas Oncology-Grapevine, Grapevine, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Texas Oncology-McAllen, McAllen, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - Texas Oncology-Midland Allison Cancer Center, Midland, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Texas Oncology-Paris, Paris, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Cancer Care Centers of South Texas- Northeast, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Texas Oncology-The Woodlands, The Woodlands, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology-Waco Highway 6, Waco, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology-Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialists-Fairfax, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Peninsula Cancer Institute-Cancer Specialists of Tidewater, Virginia Beach, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Radiology Associates of Appleton/ThedaCare Regional Medical Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Wheaton Franciscan Healthcare-Elmbrook Memorial Hospital, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Wheaton Franciscan Healthcare-Saint Francis/Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Wheaton Franciscan Healthcare-Saint Joseph/Wauwatosa Campus, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Health Sciences North, Greater Sudbury, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM-Hotel Dieu de Montreal, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan